CLINICAL TRIAL: NCT06918002
Title: A Phase 3, Open-label, Controlled, Randomized Study of Newly Diagnosed Multiple Myeloma Treatment, Designed to Evaluate the Efficacy and Safety of the Elranatamab-lenalidomide Combination as a Replacement for Chemotherapy Followed by Autologous Stem Cell Transplant in the Consolidation Phase, and to Compare Elranatamab With Standard of Care in the Maintenance Phase
Brief Title: Elranatamab/Lenalidomide Consolidation and/or Elranatamab Maintenance Versus Standard of Care After D-VRd Induction in Transplant-eligible NDMM Patients
Acronym: ElLen
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Intergroupe Francophone du Myelome (Network)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFM 2025-01; 2024-516418-39-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-10; First posted 2025-04-09 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma, Newly Diagnosed
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; daratumumab; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- D-VRD induction, ASCT and D-VRD consolidation (arm A) (Active Comparator): Standard induction therapy with 4 cycles of D-VRd, followed by HDCT (Melphalan) + ASCT, and 2 cycles of D-VRd consolidation therapy
  Interventions: Drug: Lenalidomide (Revlimid®); Drug: Daratumumab SC (Darzalex); Procedure: Autologous Stem Cell Transplantation; Drug: Bortezomib (Velcade®); Drug: Dexamethasone
- D-VRD induction followed by elranatamab and lenalidomide consolidation (arm B) (Experimental): Standard induction therapy with 4 cycles of D-VRd, followed by elranatamab and lenalidomide consolidation therapy.
  Interventions: Drug: Elranatamab; Drug: Lenalidomide (Revlimid®); Drug: Daratumumab SC (Darzalex); Drug: Bortezomib (Velcade®); Drug: Dexamethasone
- lenalidomide maintenance (Arm C) (Active Comparator): Lenalidomide monotherapy for two years (maintenance)
  Interventions: Drug: Lenalidomide (Revlimid®)
- elranatamab maintenance (Arm D) (Experimental): Elranatamab monotherapy for two years (maintenance)
  Interventions: Drug: Elranatamab

INTERVENTIONS:
Drug: Elranatamab — Elranatamab is given to arm B patients in association with lenalidomide (for consolidation) and arm D patients in monotherapy (for maintenance) as experimental arms
  Arms: D-VRD induction followed by elranatamab and lenalidomide consolidation (arm B); elranatamab maintenance (Arm D)
Drug: Lenalidomide (Revlimid®) — In association with daratumumab, bortezomib and dexamethasone (Arm A), in association with elranatamab (Arm B), in monotherapy (Arm C)
  Arms: D-VRD induction followed by elranatamab and lenalidomide consolidation (arm B); D-VRD induction, ASCT and D-VRD consolidation (arm A); lenalidomide maintenance (Arm C)
Drug: Daratumumab SC (Darzalex) — Daratumumab is given in association with bortezomib, lenalidomide and dexamethasone in induction therapy (all patients) and consolidation arm A
  Arms: D-VRD induction followed by elranatamab and lenalidomide consolidation (arm B); D-VRD induction, ASCT and D-VRD consolidation (arm A)
Procedure: Autologous Stem Cell Transplantation — ASCT is performed in consolidation for Arm A patients after induction therapy with D-VRD
  Arms: D-VRD induction, ASCT and D-VRD consolidation (arm A)
Drug: Bortezomib (Velcade®) — Bortezomib is given in associtaion with daratumumab, lenalidomide and dexamethasone in induction (all patients) and consolidation Arm A
  Arms: D-VRD induction followed by elranatamab and lenalidomide consolidation (arm B); D-VRD induction, ASCT and D-VRD consolidation (arm A)
Drug: Dexamethasone — Dexamethasone is given in association with daratumumab, bortezomib and lenalidomide in induction (all patients) and consolidation Arm A
  Arms: D-VRD induction followed by elranatamab and lenalidomide consolidation (arm B); D-VRD induction, ASCT and D-VRD consolidation (arm A)

SUMMARY:
This study is designed as a multicenter, randomized, parallel groups, open-label, phase 3 study in subjects with untreated newly diagnoses Multiple Myeloma eligible for ASCT.

824 patients will be enrolled in this study from approximately 70 study sites.

The 2 parts in the Treatment Phase are described below.

Part 1: Induction/ASCT/Consolidation Phase (1:1 Randomization)

After the screening period, patients will be randomly allocated (1:1) to either:

* Arm A (standard of care arm): standard induction therapy with 4 cycles of D-VRd, followed by HDCT (Melphalan) + ASCT, D-VRd consolidation therapy
* Arm B (experimental arm): standard induction therapy with 4 cycles of D-VRd, followed by elranatamab and lenalidomide consolidation therapy.

Part 2: Maintenance Phase (1:1 Re-randomization) Patients will be re-randomized (1:1) and will enter the Maintenance Phase upon completion of consolidation therapy.

* Arm C (standard of care arm): lenalidomide
* Arm D (experimental arm): elranatamab

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, aged over 18.
2. Patients have provided voluntary written informed consent before performing any study-related procedure.
3. Patients with newly diagnosed multiple myeloma (NDMM) eligible for high-dose chemotherapy (melphalan) and autologous stem cell transplantation (ASCT).
4. Patients with documented symptomatic NDMM according to CRAB and/or SLIM criteria, with measurable disease as defined by:

   * Presence of ≥10% monoclonal plasma cells in the bone marrow OR presence of a biopsy-proven plasmacytoma. In addition, the patient must have ≥1 of the following myeloma defining events:

     - Hypercalcemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than upper limits of normal (ULN) or >2.75 mmol/L (>11 mg/dL).

     - Renal insufficiency: creatinine clearance < 40mL/min/1.73 m2 using CKD-EPI or serum creatinine >177 μmol/L (>2 mg/dL).

     - Anemia: hemoglobin >2 g/dL below the lower limit of normal (LLN) or hemoglobin <10 g/dL.
     * Bone lesions: ≥1 osteolytic lesion on skeletal radiography, CT or PET-CT.
     * Clonal bone marrow plasma cell percentage ≥60%.
     * Serum involved/uninvolved free light chain ratio ≥100.
     * More than 1 focal lesion (≥5 mm diameter) on MRI.
   * Measurable disease as defined by serum M-component ≥5 g/L, and/or urine M-component ≥200 mg/24 h and/or serum FLC ≥100 mg/L.
5. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤2.
6. Patients must have clinical laboratory values (within 15 days of initiating induction therapy) as follows:

   • Hemoglobin ≥7.5 g/dL (≥5 mmol/L). Prior red blood cell (RBC) transfusion or the use of recombinant human erythropoietin is permitted.

   • Absolute neutrophil count (ANC) ≥1.0 G/L (granulocyte colony stimulating factor [G-CSF] use is permitted).

   • Aspartate aminotransferase (AST) ≤3 x ULN.

   • Alanine aminotransferase (ALT) ≤ 3 x ULN.

   • Total bilirubin ≤3 x ULN (except in subjects with congenital bilirubinemia, such as Gilbert syndrome, that require a direct bilirubin ≤3 x ULN).

   • Calculated creatinine clearance ≥40 mL/min/1.73 m².

   • Albumin corrected serum calcium ≤14 mg/dL (<3.5 mmol/L); or free-ionized calcium ≤6.5 mg/dL (≤1.6 mmol/L).

   • Platelet count ≥50 Giga/L for subjects who have <50% of bone marrow nucleated cells as plasma cells. If not, platelet count >30 G/L (platelets transfusions done during the 15 days before initiating induction therapy are not permitted).
7. Women of childbearing potential must have a negative serum or urine pregnancy test during the screening period before randomization AND within 3 days before of initiating induction therapy.

Exclusion Criteria:

1. Subjects previously treated with any systemic therapy for multiple myeloma. Patients are allowed corticosteroids during screening not >160 mg of dexamethasone (or equivalent). Patients with concurrent radiotherapy (localized) within the 14 days before initiating induction therapy are not eligible (If possible, in these cases, enrolment should be deferred).
2. Subject with ongoing Grade ≥ 3 peripheral sensory or motor neuropathy.
3. Subject with history of GBS or GBS variants, or history of any Grade ≥3 peripheral motor polyneuropathy.
4. Subject with a current diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance, smoldering multiple myeloma, or solitary plasmacytoma.
5. Subject has a diagnosis of Waldenström's macroglobulinemia, or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions.
6. The subject has had plasmapheresis within 14 days of initiating induction therapy.
7. Subject with clinical signs of meningeal involvement of multiple myeloma.
8. The subject has plasma cell leukemia (by WHO criterion: ≥5% of plasma cells in the peripheral blood) or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
9. Subject has any concurrent medical or psychiatric condition or disease (e.g., active systemic infection, uncontrolled diabetes, acute diffuse infiltrative pulmonary disease) that is likely to interfere with the study procedures or results, or that in the opinion of the investigator, would constitute a hazard for participating in this study.
10. Subject has clinically significant cardiac disease, including:

    • Subject has had myocardial infarction within 1 year before initiating induction therapy, or currently has an unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association [NYHA] class III IV).

    • Subject has uncontrolled cardiac arrhythmia (common terminology criteria for adverse events [CTCAE] version 4 grade ≥2) or clinically significant electrocardiography (ECG) abnormalities.

    • Subject with a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec (12-lead ECG).
11. Subjects taking systemic treatment with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort (millepertuis) within the 14 days before initiating induction therapy.
12. Known intolerance to steroids, mannitol, pregelatinized starch, sodium stearyl fumarate, histidine (as base and hydrochloride salt), arginine hydrochloride, poloxamer 188, sucrose or any of the other components of study intervention that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents.
13. Known allergies to any of the study medications, their analogues, or excipients in the various formulations.
14. Subjects who have had major surgery within 2 weeks before study inclusion (signing of the informed consent) OR will not have fully recovered from surgery before initiating induction therapy OR have surgery planned during their study participation. Kyphoplasty and vertebroplasty are not considered as major surgery.
15. Subjects with any prior or concurrent invasive malignancy (other than multiple myeloma) within 10 years of study inclusion study, except for adequately treated basal cell or squamous cell carcinoma of the skin, in situ carcinoma of the cervix, or localized prostate adenocarcinoma diagnosed ≥3 years ago and without evidence of biological failure, or other cancers for which the subject has undergone potentially curative therapy and has without evidence of relapse/recurrence for ≥10 years.
16. Pregnant or breast-feeding women.

Women that refuse to abstain from heterosexual intercourse or refuse to use adequate contraceptives during heterosexual intercourse starting at least 4 weeks before initiating induction therapy and continually until at least 4 weeks after discontinuing lenalidomide,90 days after discontinuing daratumumab and 6 months after discontinuing elranatamab.

18. Men with partners of childbearing potential, even men with a successful vasectomy, that refuse to use a condom during intercourse, from initiating induction therapy to ≥4 weeks ys after discontinuing lenalidomide,. Furthermore, men must agree to not donate sperm during this period.

19. Known positive for HIV or active hepatitis A, B or C: Uncontrolled or active HBV infection: Patients with positive HBsAg and/or HBV DNA

Of note:

Patients can be eligible if anti-HBc IgG positive (with or without positive anti-HBs) but HBsAg and HBV DNA are negative.

o If anti-HBV therapy in relation to prior infection was started before initiation of IMP, the anti-HBV therapy and monitoring should continue throughout the study treatment period.

Patients with negative HBsAg and positive HBV DNA observed during screening period will be evaluated by a specialist for start of anti-viral treatment: study treatment could be proposed if HBV DNA becomes negative, and all the other study criteria are still met.

* Active HCV infection: positive HCV RNA and negative anti-HCV.

Of note:

Patients with antiviral therapy for HCV started before initiation of IMP and positive HCV antibodies are eligible. The antiviral therapy for HCV should continue throughout the treatment period until seroconversion.

Patients with positive anti-HCV and undetectable HCV RNA without antiviral therapy for HCV are eligible.

20. Patient with an active systemic infection or severe infections requiring parenteral administration of antibiotics.

21. Patients with a gastrointestinal disease/disorder that may significantly impact the absorption of oral treatments.

22. Patients unable or unwilling to undergo antithrombic prophylaxis.

23. A person under guardianship, trusteeship, or deprived of freedom by a judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 824 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2036-05 (Estimated); Study Completion 2036-05 (Estimated)

PRIMARY OUTCOMES:
Part 1 (induction/consolidation) from Randomization 1 (R1): to assess whether consolidation therapy with elranatamab and lenalidomide is superior to standard of care, in terms of Minimal Residual Disease (MRD) negativity rate | at end of consolidation, up to 36 months
  To assess whether consolidation therapy with elranatamab and lenalidomide is superior to standard of care, in terms of MRD negativity rate.
Part 2 (maintenance) from Randomization 2 (R2): to assess whether maintenance therapy with elranatamab is superior to standard of care, in terms of Progression Free Survival (PFS). | from the date of second randomization to the date of confirmed PD (IMWG criteria,) or death from any cause, whichever came first, assessed up to 93 monts
  To assess whether maintenance therapy with elranatamab is superior to standard of care, in terms of PFS.
Key secondary objectives: Part 1 (induction/consolidation) from R1: to assess whether consolidation therapy with elranatamab and lenalidomide is superior, in terms of PFS | PFS defined as the time interval from the date of first randomization to the date of confirmed Progression Disease (IMWG criteria) or death from any cause, whichever occurs first., assessed up to 128 months
  To assess whether consolidation therapy with elranatamab and lenalidomide is superior, in terms of PFS
Key secondary objectives: Part I (induction/consolidation) from R1: to assess whether consolidation therapy with elranatamab and lenalidomide is superior to standard of care, in terms of Overal Survival (OS) | up to 128 months
  To assess whether consolidation therapy with elranatamab and lenalidomide is superior to standard of care, in terms of OS

SECONDARY OUTCOMES:
Part 1 (induction/consolidation) from R1: to assess the efficacy of consolidation therapy with elranatamab and lenalidomide compared to standard of care | End of consolidation phase, up to 36 months
  To assess the efficacy of consolidation therapy with elranatamab and lenalidomide compared to standard of care: Overall response rate (ORR), Very good partial response (VGPR) rate, Complete response (CR) rate
Part 2 (maintenance) from R2: to assess the efficacy of maintenance therapy with elranatamab | end of maintenance, up to 58 months
  To assess the efficacy of maintenance therapy with elranatamab:
  * Overall response rate (ORR) in maintenance
  * Very good partial response (VGPR) rate in maintenance
  * Complete response (CR) rate in maintenance
assess safety & Tolerability during induction, and during consolidation and maintenance therapy: Adverse events (AE), serious Adrverse events (SAE) and And adverse events of special interest (AESI) rates - Incidence of Treatment-Emergent Adverse Events | through study completion, up to 128 months
  To assess safety during induction, and during consolidation and maintenance therapy: AEs, SAE and AESI rates , Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Throughout the study to evaluate the impact of treatment on health-related Quality of Life (QoL) using Rework questionnaire | through study completion, up to 128 months
  To evaluate the impact of treatment on health-related QoL: Rework questionnaire
Part 2 (maintenance) from Randomization 2 (R2): to assess the efficacy of maintenance therapy with elranatamab, Progression Free Survival 2 form Randomization 2 | up to 128 months
  To assess the efficacy of maintenance therapy with elranatamab:
  - PFS of subsequent/next treatment line (PFS2 from R2)
Part 2 (maintenance) from R2: to assess the efficacy of maintenance therapy with elranatamab, in term of Minimal Residual Disease negativity | 12 months post R2, up to 71 months
  To assess the efficacy of maintenance therapy with elranatamab:
  - MRD negativity at 12 months post R2
Throughout the study: to evaluate the impact of treatment on health-related Quality of Life (QoL) using EQ-5D-5L | Though study completion, an average of 11 years
  To evaluate the impact of treatment on health-related QoL: scale title :EQ-5D-5L , the minimum value is 0 and maximum value is 100 (100 corresponds to the best health that patient can imagine, 0 corresponds to the worst health that patient can imagine
Part 2 (maintenance) from R2: To assess the efficacy of maintenance therapy with elranatamab (OS R2) | up to 128 months
  To assess the efficacy of maintenance therapy with elranatamab:
  - Overall survival from second randomization (OS R2)

OTHER OUTCOMES:
EXPLORATORY OBJECTIVES: to assess the impact of genomic markers (from Next generation sequencing (NGS) and Whole Genome Sequencing (WGS)) on outcome | up to 128 months
  To assess the impact of genomic markers (from NGS and WGS) on outcome: MRD negativity rate as determined by NGS with a sensitivity of at least 10-5 - PFS1 and OS
EXPLORATORY OBJECTIVES: to assess Immune mechanisms predicting Elra-Len vs ASCT efficacy | up to 128 months
  Impact of the microenvironment (Immune mechanisms predicting Elra-Len vs ASCT efficacy) according to outcome (MRD, PFS and OS) rates
EXPLORATORY OBJECTIVES: to assess the impact of PET imaging parameters/variables on outcome | End of consolidation phase, up to 36 months
  rate of PET imaging positive / negative according to outcome (MRD, PFS and OS) rates
EXPLORATORY OBJECTIVES: To determine influence of M-component measurement assessed by mass spectrometry on outcome | up to 128 months
  To determine influence of M-component measurement assessed by mass spectrometry on outcome
EXPLORATORY OBJECTIVES: To determine influence of circulating tumor cells on outcome in term of PFS1 and OS | up to 128 months
  To determine influence of circulating tumor cells on outcome in term of PFS1 and OS

CONTACTS AND LOCATIONS:
Overall Officials: Chanaz LOUNI, Study Director — The Institute for Functional Medicine; Aurore PERROT, Prof, Principal Investigator — IUCT Toulouse France; Cyrille TOUZEAU, Prof, Principal Investigator — CHU Nantes France
Locations (64):
- France (64):
  - Amiens, Amiens
  - CHU Angers, Angers
  - Ch Annecy Genevois, Annecy
  - Centre Hospitalier d'Argenteuil Victor Dupouy, Argenteuil
  - Centre Hospitalier H. Duffaut, Avignon
  - Centre hospitalier de la Côte Basque, Bayonne
  - CHU Besançon, Besançon
  - Centre Hospitalier Simone Veil, Blois
  - Hôpital Avicenne, Bobigny
  - CHU Bordeaux - Hopital Haut Lévêque - Centre F. Magendi, Bordeaux
  - CH Fleyriat, Bourg-en-Bresse
  - CHRU Brest - Hôpital A. Morvan, Brest
  - CHU Caen - Côte de Nacre, Caen
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - CHMS Centre Hospitalier Métropole Savoie, Chambéry
  - Hopital Louis Pasteur, Chartres
  - Hôpital d'Instruction des Armées Percy, Clamart
  - Chu Estaing, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CHU Henri Mondor, Créteil
  - CHU Dijon, Dijon
  - Institut de cancérologie de Bourgogne, Dijon
  - Centre Hospitalier de Dunkerque, Dunkirk
  - CHU de Grenoble, Grenoble
  - CHU de la Réunion Site SUD (Terre Sainte), La Réunion
  - CHD Vendée, La Roche-sur-Yon
  - Hopital Monod, Le Havre
  - CH Le mans, Le Mans
  - CHRU Hôpital Claude Huriez, Lille
  - Centre Hospitalier Universitaire (CHU) de Limoges, Limoges
  - Centre Hospitalier Lyon Sud, Lyon
  - Grand Hopital Est Francilien (GHEF) Site de Meaux, Meaux
  - Hôpital de Mercy (CHR Metz-Thionville), Metz
  - Centre de Recherche Clinique / GHT des Landes, Mont-de-Marsan
  - Hopital Saint Eloi - CHU Montpellier, Montpellier
  - Hôpital E. Muller, Mulhouse
  - CHRU Hôpitaux de Brabois, Nancy
  - CHRU Hôtel Dieu, Nantes
  - Hôpital Archet 1, Nice
  - CHU Carémeau, Institut de Cancérologie du Guard, Nîmes
  - CHR Orléans, Orléans
  - CHU Hôpital Saint Antoine, Paris
  - Hôpital Cochin, Paris
  - Hôpital Necker, Paris
  - Hôpital Saint Louis, Paris
  - La Pitié Salpêtrière, Paris
  - CH Saint Jean, Perpignan
  - Centre Hospitalier de Perigueux, Périgueux
  - CHU Poitiers - Pôle régional de Cancérologie, Poitiers
  - Centre hospitalier René Dubost, Pontoise
  - Centre Hospitalier de Quimper Cornouaille, Quimper
  - Hôpital Robert Debré, Reims
  - CHRU Hôpital de Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier Saint Brieuc, Saint-Brieuc
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest
  - Centre Hospitalier de Saint-Quentin, Saint-Quentin
  - CHU Strasbourg, Strasbourg
  - Centre hospitalier, Tarbes
  - Pôle IUCT Oncopole CHU, Toulouse
  - CHRU Hôpital Bretonneau - Centre Henry Kaplan, Tours
  - CH Bretagne Atlantique Vannes et Auray - P. Chubert, Vannes
  - CHV André Mignot - Université de Versailles, Versailles
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No